CLINICAL TRIAL: NCT02966379
Title: Hearing Preservation and Electro-acoustic Stimulation With EVO® Electrode Lead and Zebra® Sound Processor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIC_06
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Cochlear Implant
Keywords: Electroacoustic stimulation
MeSH Terms: interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear implantation (Experimental): Cochlear implantation with EVO electrode lead. This electrode lead has been specially designed for atraumatic surgery, in order to preserve the residual hearing of the patients included in the study. All patients are implanted with the same electrode lead.
  Interventions: Device: cochlear implantation

INTERVENTIONS:
Device: cochlear implantation — Surgery is standardized in order to have the same procedure for all patients and to preserve a maximum of residual hearing:
  * Corticosteroïds (1mg/kg solumedrol) at anesthetic induction ,
  * mastoidectomy + posterieur tympanostomy ,
  * insertion through round window,
  * stop at the first resistance point

SUMMARY:
Some candidates to cochlear implantation can have residual low frequencies hearing. The EVO electrode lead has been specifically designed to preserve this residual hearing through surgery. It is then possible to provide the patient with a electro-acoustic stimulation (EAS) which combines both an acoustical stimulation for the preserved low frequency hearing and an electrical stimulation through the cochlear implant. The major aim of this study is to evaluate hearing preservation after implantation with the EVO electrode lead.

The secondary outcome is to evaluate the benefit of EAS stimulation provided by the Zebra speech processor.

DETAILED DESCRIPTION:
Some candidates to cochlear implantation can have residual low frequencies hearing. The EVO electrode lead has been specifically designed to preserve this residual hearing through surgery. It is then possible to provide the patient with a electro-acoustic stimulation (EAS) which combines both an acoustical stimulation for the preserved low frequency hearing and an electrical stimulation through the cochlear implant. Literature showed the EAS stimulation can lead to better speech understanding, especially in noisy situation, and can provide important information about intonating or melodic contours, thus increasing sound quality and music perception.

Objectives The major aim of this study is to evaluate hearing preservation after implantation with the EVO electrode lead.

The secondary outcome is to evaluate the benefit of EAS stimulation provided by the Zebra speech processor.

Methods Unaided tonal audiograms are measured for cochlear implant candidates with low frequency residual hearing before and after cochlear implantation with the EVO electrode lead.

Aided tonal audiograms and speech intelligibility in quiet and in noise are measured after implantation with the three modes of stimulation (acoustic stimulation AS, electric stimulation ES, and electro-acoustic stimulation EAS).

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate
* Above 18 years old
* Candidate for cochlear implantation
* Residual hearing in low frequencies (auditory thresholds better than or equal to 70 dB up to 500 Hz
* Native or fluent French speaker

Exclusion Criteria:

* No affiliation to social security
* No agreement
* Vulnerable patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Change in pure tone audiometric thresholds at 125, 250, 500, 750, 1000, 2000 and 4000 Hz between pre and post implantation | 2 weeks pre-implantation, 1 month post-implantation, 1, 3, 6 and 12 months post-activation
  Change from pre-implantation pure tone audiometric thresholds at 125, 250, 500, 750, 1000, 2000 and 4000 Hz at 1 month post implantation with the EVO electrode lead and at 1, 3, 6 and 12 months post-activation

SECONDARY OUTCOMES:
Percentage of words and phonemes correctly identify with "Les listes cochléaires de Lafon" presented in quiet with the speech processor providing acoustic stimulation (AS), Electric Stimulation (ES) or electro-acoustic stimulation (EAS). | 3, 6 and 12 months post activation
  Percentage of words and phonemes correctly identify with "Les listes cochléaires de Lafon" when presented in quiet with the three modes of stimulation (AS, ES and EAS). Speech understanding is evaluated at 3, 6 and 12 months post activation
Percentage of words and phonemes correctly identify with "Les listes cochléaires de Lafon" presented in cocktail party noise with the speech processor providing acoustic stimulation (AS), Electric Stimulation (ES) or electro-acoustic stimulation (EAS). | 3, 6 and 12 months post activation
  Percentage of words and phonemes correctly identify with "Les listes cochléaires de Lafon" when presented in cocktail party noise at 0 and +10 dB Speech to Noise Ratio (SNR) with the three modes of stimulation (AS, ES and EAS). Speech understanding is evaluated at 3, 6 and 12 months post activation
Quality of life questionnaire. Evaluation of satisfaction on a scale from 0 (unsatisfactory) to 10 (satisfactory) of everyday life listening situations. | 2 weeks pre op, 3, 6 and 12 months post-activation
Intonation perception task measuring the JND (just noticeable difference) in frequency necessary to discriminate two sounds | 6 and 12 months post activation
Surgery questionnaire evaluating the surgical technique, the presence of problems during surgery, the quality of insertion and surgeon satisfaction with multiple choice questions, close questions and scales from 0 to 10. | single evaluation at implantation only
  Surgery questionnaire evaluating the surgical technique (multiple choice questions), the presence of problems during surgery (multiple choice questions), the difficulty of insertion of the implant (scales from 0 - impossible to 5 - very easy; or 0 -very easy to 5 - impossible on inverted questions), the tools used for the insertion (multiple choice questions), the duration of insertion (secondes or minutes),the number of electrode inserted, the number of attempts to insert, and surgeon satisfaction (multiple choice questions between "easy", "medium" and "difficult")

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gnansia, Dr, Study Director — Oticon Medical; Yann NGUYEN, Dr, Principal Investigator — APHP Pitie salpetriere
Locations (8):
- France (8):
  - CHU Bordeaux Pellegrin, Bordeaux
  - CHRU Lille Hôpital Roger Salengro, Lille
  - CHU Lyon Hôpital Edouard Herriot, Lyon
  - APHM - Hôpital Nord Marseille, Marseille
  - CHRU de Nancy hôpital Central, Nancy
  - IUFC - CHU Nice, Nice
  - APHP Pitie salpetriere, Paris
  - CHU Rennes Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No